CLINICAL TRIAL: NCT01820312
Title: A Phase II Study to Evaluate Low-Dose Fractionated Radiotherapy (LDFRT) and Chemotherapy in Recurrent and Inoperable Squamous Cell Carcinoma (SCC) of the Head and Neck After Radiotherapy Failure
Brief Title: A Phase II Study to Evaluate Low-Dose Fractionated Radiotherapy (LDFRT)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to no enrollment.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 136191
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Low-Dose Fractionated Radiation Therapy/Paclitaxel

SUMMARY:
The purpose of this study is to determine if low-dose radiation therapy and the chemotherapy drug paclitaxel is effective in treating head and neck cancer that has returned after treatment with standard radiation therapy alone, but cannot be removed by surgery. The overall total dose received of both the chemotherapy and radiation therapy will be less than that typically given as standard of care; however, the Food and Drug Administration (FDA) has not evaluated the safety and effectiveness of this combination therapy. In addition, this study will gather information about the effects of radiation therapy and chemotherapy on subject's overall quality of life.

DETAILED DESCRIPTION:
This study will evaluate a combination therapy of paclitaxel and LDFRT. The paclitaxel will be commercially available drug product dispensed by a licensed pharmacist at UAMS. Radiotherapy will be delivered using either the TomoTherapy Treatment System (TomoTherapy, Inc.) or the Varian High Energy Linear Accelerator (Varian Medical Systems).

Subjects will undergo CT imaging (to include neck, chest, abdomen and pelvis) as part of the standard of care approximately 7 to 21 days prior to initiation of this therapy. Additional CT imaging will be done at UAMS approximately 3 months after completion of protocol therapy and every 3 months subsequently until progression or completion of the study whichever comes first. These CT imaging's will be obtained for recurrent tumor evaluation and determination of the presence or absence of distant metastasis, as part of the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject 18 years of age and older, male or female, of all races and ethnicities.
2. Subject with prior histologically confirmed advanced squamous-cell carcinoma of the head and neck that failed prior traditional chemoradiotherapy with at least a 3-month disease-free interval from the completion of the initial curative treatment.
3. Recurrence must have been confirmed via biopsy.
4. Subject must have an ECOG performance status of 0, 1 or 2.
5. Has undergone CT imaging within 21 days prior to treatment as part of routine care.
6. Measurable disease by CT.
7. Subject deemed likely to survive for at least 6 months.
8. Subject is able and willing to provide written informed consent to participate in the study.
9. If the subject is a female of childbearing age, the subject should have a negative urine pregnancy test and be practicing strict birth control (estrogen-containing oral contraceptives or an intrauterine device) throughout the study and for 3 months after completion of protocol treatment. Women who have had a hysterectomy are exempt from these requirements. This is routine for any patient undergoing treatment.
10. History of laboratory criteria as specified below (within 21 days prior to enrollment) Hemoglobin ≥ 9 g/dl Platelet count >100,000 per microliter CO2 (carbon dioxide): 22-32 meq/L Creatinine: < 1.5 mg/dL or eGFR>40 ml/min Serum bilirubin <1.6 mg/dl. White blood count > 3,000 per microliter or ANC > 1500 per microliter Serum calcium <10.5 mg/dl.

Exclusion Criteria:

1. The tumor is not clearly shown on diagnostic imaging studies
2. Subject is pregnant.
3. Subject with known allergies/hypersensitivity to paclitaxel.
4. Subjects with poor renal function as demonstrated by serum creatinine (>1.5 mg/dl) and EGFR <40 mL/min, which would preclude the using of image contrast agents.
5. Subject with a planned surgical procedure within the next 30 days.
6. Subject has distant metastasis (with the exception of single stable distant metastasis that does not decrease life expectancy to less than 6 months).
7. Subject is of childbearing potential and will not use adequate contraceptive protection.
8. Subject who is breastfeeding.
9. Subject of childbearing potential who has a positive (+) urine pregnancy test.
10. Subject has received treatment with an experimental drug or entered another clinical trial within the prior 30 days.
11. Subject has received radiotherapy to the head and neck region within the prior 3 months.
12. Subject is not willing or able to complete the visit requirements of this protocol.
13. Peripheral neuropathy of any etiology.
14. Any other condition that the PI feels will be an endangerment to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Objective Response (OR) | OR will be determined in each subject 3 months following therapy using CT imaging performed for clinical-care purposes
  Objective Response (OR). OR will be defined according to RECIST v1.1 criteria as either a complete or partial response. OR will be determined in each subject 3 months following therapy using CT imaging performed for clinical-care purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Penagaricano, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rick, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No